CLINICAL TRIAL: NCT00475111
Title: Stress and Adaptation in Rheumatoid Arthritis (SARA)
Brief Title: Cognitive Behavioral Therapy Treatments for Adults With Rheumatoid Arthritis (The SARA Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Arthritis Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AR041687 (NIH); R01AR041687 (NIH)
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Cognitive Behavioral Intervention; Emotion Regulation; Pain Management; Psychological Adaptation; Coping Efficacy; Markers of Disease Activity
MeSH Terms: conditions — Arthritis, Rheumatoid; Emotional Regulation; Agnosia | interventions — Cognitive Behavioral Therapy; Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): People in Group 1 will participate in CBT for Pain (CBT-P), which will focus on altering thought processes as a way to cope more effectively with pain.
  Interventions: Behavioral: Cognitive Behavior Therapy for Pain (CBT-P)
- 2 (Experimental): People in Group 2 will participate in Mindfulness Medication for Emotion Regulation (MM-ER), a type of CBT that focuses on being more aware of one's emotions and regulating them.
  Interventions: Behavioral: Mindfulness Meditation for Emotion Regulation (MM-ER)
- 3 (Experimental): Group 3 participants will serve as controls and receive educational information on the causes of, course of, and treatment for RA.
  Interventions: Behavioral: Rheumatoid arthritis education

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy for Pain (CBT-P)
  Arms: 1
Behavioral: Mindfulness Meditation for Emotion Regulation (MM-ER)
  Arms: 2
Behavioral: Rheumatoid arthritis education
  Arms: 3

SUMMARY:
Rheumatoid arthritis (RA) is an autoimmune disease that causes long-term inflammation of the joints and occasionally, other body tissues. The purpose of this study is to evaluate two different types of cognitive behavioral therapy (CBT) in reducing RA disease activity and improving mental health of adults with RA.

DETAILED DESCRIPTION:
Symptoms of RA include swelling, pain, stiffness, and redness in the joints. Over time, joint deformity, joint destruction, and loss of function can occur. Even simple tasks of daily living can become difficult to manage for people with RA. Current treatment aims to improve symptoms, but there is currently no cure for the disease. Dealing with the long-term pain and the unpredictability of RA can cause symptoms of depression, which is common among people with RA, especially early in the disease. Improving coping skills and minimizing emotional stress may help improve the overall health of people with RA. CBT is a form of psychotherapy that emphasizes the important role of thinking in how we feel and what we do. This type of therapy emphasizes that people can change the way they think to feel or act better even if the situation does not change. The purpose of this study is to evaluate two different types of CBT that focus on stress, pain, and depression responses in reducing disease activity and improving mental health of adults with RA.

This study will last about 15 months. Initially, all participants will fill out a diary report about their symptoms for a total of 30 days. Half of the study participants will undergo a 2- to 3-hour lab session that will include blood collection, vital signs measurements, joint exams, questionnaires, and an interview about symptoms and medical history. All participants will then be randomly assigned to one of the following three groups:

* People in Group 1 will participate in CBT for Pain (CBT-P), which will focus on altering thought processes as a way to cope more effectively with pain.
* People in Group 2 will participate in Mindfulness Medication for Emotion Regulation (MM-ER), a type of CBT that focuses on being more aware of one's emotions and regulating them.
* Group 3 participants will serve as controls and receive educational information on the causes of, course of, and treatment for RA.

Participants in all three groups will attend 2-hour weekly sessions of their treatment for 8 weeks. After treatment, all participants will undergo a 2- to 3-hour lab session that will include blood collection, vital signs measurements, joint exams, questionnaires, and an interview about symptoms and medical history. Participants will also fill out another daily diary report about their symptoms for 30 days. A follow-up questionnaire will be mailed to participants 6 months following the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA

Exclusion Criteria:

* Currently taking cyclical estrogen replacement therapy
* Diagnosis of lupus

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2001-03; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Pain, physical functioning, coping efficacy, positive and negative emotional affect, and depression | 6 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alex J. Zautra, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Tempe, Arizona, United States

REFERENCES:
- [Background] Conner TS, Tennen H, Zautra AJ, Affleck G, Armeli S, Fifield J. Coping with rheumatoid arthritis pain in daily life: within-person analyses reveal hidden vulnerability for the formerly depressed. Pain. 2006 Dec 15;126(1-3):198-209. doi: 10.1016/j.pain.2006.06.033. Epub 2006 Aug 14. PMID 16904829
- [Background] Davis MC, Affleck G, Zautra AJ, Tennen H. Daily interpersonal events in pain patients: applying action theory to chronic illness. J Clin Psychol. 2006 Sep;62(9):1097-113. doi: 10.1002/jclp.20297. PMID 16810668
- [Background] Zautra AJ, Affleck GG, Tennen H, Reich JW, Davis MC. Dynamic approaches to emotions and stress in everyday life: Bolger and Zuckerman reloaded with positive as well as negative affects. J Pers. 2005 Dec;73(6):1511-38. doi: 10.1111/j.0022-3506.2005.00357.x. PMID 16274444
- [Background] Zautra AJ, Fasman R, Parish BP, Davis MC. Daily fatigue in women with osteoarthritis, rheumatoid arthritis, and fibromyalgia. Pain. 2007 Mar;128(1-2):128-35. doi: 10.1016/j.pain.2006.09.004. Epub 2006 Oct 20. PMID 17055648
- [Derived] Davis MC, Zautra AJ, Wolf LD, Tennen H, Yeung EW. Mindfulness and cognitive-behavioral interventions for chronic pain: differential effects on daily pain reactivity and stress reactivity. J Consult Clin Psychol. 2015 Feb;83(1):24-35. doi: 10.1037/a0038200. Epub 2014 Nov 3. PMID 25365778
- [Derived] Zautra AJ, Davis MC, Reich JW, Nicassario P, Tennen H, Finan P, Kratz A, Parrish B, Irwin MR. Comparison of cognitive behavioral and mindfulness meditation interventions on adaptation to rheumatoid arthritis for patients with and without history of recurrent depression. J Consult Clin Psychol. 2008 Jun;76(3):408-421. doi: 10.1037/0022-006X.76.3.408. PMID 18540734
- See also: Click here for the Stress and Adaptation in Rheumatoid Arthritis (SARA) study's intervention manuals — http://www.public.asu.edu/~atajz/